CLINICAL TRIAL: NCT00054288
Title: Escalating Irinotecan (CPT-11) Administered 24 Hours Prior To Gemcitabine In Patients With Refractory Solid Tumors
Brief Title: Irinotecan and Gemcitabine in Treating Patients With Refractory Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Nithya Ramnath, MD, Roswell Park Cancer Institute
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270343; RPCI-DS-01-18
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining irinotecan with gemcitabine in treating patients who have refractory advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of irinotecan when administered with gemcitabine in patients with refractory advanced solid tumors.
* Determine the antitumor activity and toxicity of this regimen in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this regimen in these patients.
* Determine the optimal dose and time interval for this regimen in these patients.

OUTLINE: This is an open-label, non-randomized, dose-escalation study of irinotecan.

Patients receive irinotecan IV over 90 minutes on days 1 and 8 and gemcitabine IV over 30 minutes on days 2 and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor that is refractory to prior treatment

  * Considered incurable with other modalities
* Measurable or evaluable disease

  * The following are not considered measurable or evaluable:

    * Bone metastases
    * Pleural, pericardial, or peritoneal effusions
    * Irradiated lesions (unless progression is documented after radiotherapy)
  * Metastatic disease that has been followed using serum tumor markers allowed
* No symptomatic brain metastases
* Brain metastases may not be sole site of metastatic disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* AST and ALT no greater than 1.5 times normal
* Bilirubin no greater than 1.5 mg/dL
* No clinically apparent jaundice

Renal

* Creatinine no greater than 1.6 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* Cardiac function normal
* No uncontrolled heart disease
* No myocardial infarction within the past 3 months
* No congestive heart failure
* No unstable or uncontrolled angina

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection requiring systemic therapy
* No uncontrolled seizures
* No uncontrolled diabetes mellitus

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior gemcitabine
* No prior camptothecin compounds
* Prior irinotecan allowed
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 14 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior clinical trial participation
* No other concurrent investigational medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-08; Primary Completion 2003-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States